CLINICAL TRIAL: NCT03069677
Title: Music vs Midazolam During Preoperative Nerve Block Placement: A Prospective, Randomized Controlled Study
Brief Title: Music vs Midazolam During Preop Nerve Block Placement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 826754
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Results first posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Anxiety; Peripheral Nerve Block
Keywords: midazolam
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy; Midazolam

STUDY DESIGN:
Intervention Model Description: 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Music group (Active Comparator): research-selected music
  Interventions: Other: music
- Midazolam group (Active Comparator): IV midazolam (1mg to 2mg max)
  Interventions: Drug: Midazolam

INTERVENTIONS:
Other: music — patients in this group will receive research-selected music after the golden moment has been completed between the patient, provider, and nursing staff
  Arms: Music group
Drug: Midazolam — patients in this group will receive IV midazolam (1mg to 2mg max) after the golden moment has been completed
  Other Names: Hypnovel
  Arms: Midazolam group

SUMMARY:
The purpose of this study is to determine if there are differences in anxiety scores, heart rate, blood pressure, and oxygen status when using sedation medication versus music while undergoing a peripheral nerve block before your surgery.

DETAILED DESCRIPTION:
The general flow of the study will be conducted as follows:

1. Research coordinator will call or approach patients who are scheduled for a surgical procedure that is planning for a peripheral nerve block either for the primary anesthetic or for postoperative pain control to be placed in the preoperative bay in the ambulatory surgical center.
2. Research coordinator will discuss the purpose of our study and explain the study in detail for the patient. If a patient agrees to participate, then we will have the patient sign the informed consent for the study. If patient is on the phone and decides to participate, the patient will sign the informed consent upon arriving to Penn Medicine University City (PMUC).
3. Once the patient signs the informed consent for the peripheral nerve block by anesthesia team. The patient randomized will be revealed to either music or IV midazolam. The pre-procedure anxiety score will then be obtained using the STAI-6 validated tool.
4. The golden moment will be conducted between the patient, provider, and nursing staff. Once this golden moment is completed, the anxiolytic intervention will start (music or IV midazolam)*
5. The preoperative nerve block will be conducted by the regional anesthesia block team.
6. Once the nerve block is complete, we will obtain the post-procedure anxiety score using the STAI-6 validated tool.
7. Once the post-procedure anxiety score has been obtained, we will also obtain the patient satisfaction score, the provider satisfaction score, and the evaluation of any difficulties in communication between the provider and patient. After these questions have been obtained, the study is complete.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are >18 years of age, who will give informed consent in receiving a peripheral nerve block in the preoperative bay for their primary anesthetic and/or for their postoperative pain control.

Exclusion Criteria:

* significant psychiatric disorder such as generalized anxiety disorder, panic disorder, depression, psychosis, bipolar disorder; individuals who were incompetent to give informed consent; pregnant and/or breast feeding patients; any underlying coagulopathy, infection or other factors which would be a contraindication to receiving a peripheral nerve block; hypersensitivity to midazolam; and history of renal impairment. Patients who were extremely anxious (scores 50 and greater on the State Trait Anxiety Inventory-6 (STAI-6) tool) were also excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2018-05-11 (Actual); Study Completion 2018-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veena Graff, MD, MS, Principal Investigator — University of Pennsylvania, Anesthesia
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Graff V, Cai L, Badiola I, Elkassabany NM. Music versus midazolam during preoperative nerve block placements: a prospective randomized controlled study. Reg Anesth Pain Med. 2019 Jul 18:rapm-2018-100251. doi: 10.1136/rapm-2018-100251. Online ahead of print. PMID 31320504

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Music Group | Midazolam Group
Started | 80 | 80
Completed | 77 | 77
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Population: there was incomplete collection of data and patients dropped out which resulted in 77 total analyzed participants in this group
Groups:
- Total: Total of all reporting groups
Arm/Group | Music Group | Midazolam Group | Total
Number analyzed (Participants) | 77 | 80 | 157
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 77 | 80 | 157
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (15.6) | 46 (16) | 45.5 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 50 | 102
  Male | 25 | 30 | 55
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 52 | 50 | 102
  Race: Black | 21 | 23 | 44
  Race: Asian | 4 | 5 | 9
  Race: Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Anxiety Levels
Description: Spielberger State-Trait Anxiety Inventory 6
  Scale range is from 20 to 80. Higher the score, the higher the anxiety level is.
Time Frame: 1-2 minutes before conducting golden moment for nerve block placement and immediately after nerve block placement (less than 1 minute after)
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Music Group | Midazolam Group
Number analyzed (Participants) | 77 | 80
score on a scale
  Pre-STAI-6 Scores | 33.3 [23.3 to 41.7] | 30 [20 to 40]
  Post-STAI-6 Scores | 30 [20 to 40] | 23.3 [20 to 33.3]

2. Primary Outcome: Change in STAI-6 Scores From Post to Pre.
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Music Group | Midazolam Group
Number analyzed (Participants) | 77 | 80
score on a scale | -1.6 (10.7) | -4.2 (11)

3. Secondary Outcome: Patient Satisfaction Scores of the Experience During Procedure
Description: survey which assess satisfaction on a 10-point numeric rating scale
  Scale ranges from 0 to 10. A higher number indicates a higher satisfaction
Time Frame: immediately after nerve block placement (less than 1 minute after)
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Music Group | Midazolam Group
Number analyzed (Participants) | 77 | 80
units on a scale | 8 [5 to 9] | 9 [7 to 10]

4. Secondary Outcome: Provider Satisfaction Scores of the Experience During Procedure
Description: as for outcome 3
Time Frame: immediately after nerve block placement (less than 1 minute after)
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Music Group | Midazolam Group
Number analyzed (Participants) | 77 | 80
units on a scale | 9 [8 to 10] | 10 [8 to 10]

5. Secondary Outcome: Evaluation of Difficulties in Communication From Provider to Patient and Patient to Provider
Description: surveyed on a 5-point Likert scale
  Scale ranges from 1 to 5; the higher the number, the more difficult it is to communicate.
Time Frame: immediately after nerve block placement (less than 1 minute after)
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Music Group | Midazolam Group
Number analyzed (Participants) | 77 | 80
score on a scale
  Patient Perspective on Communication | 1 [1 to 2] | 1 [1 to 1]
  Physician Perspective on Communication | 1 [1 to 2] | 1 [1 to 1]

6. Secondary Outcome: Block Times
Description: differences amongst music and midaz group
Time Frame: immediately after nerve block placement (less than 1 minute after)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Music Group | Midazolam Group
Number analyzed (Participants) | 77 | 80
minutes | 6.7 (4.2) | 7 (4.2)

ADVERSE EVENTS:
Time Frame: one year
Groups:
- Music Group: research-selected music
  music: patients in this group will receive research-selected music after the golden moment has been completed between the patient, provider, and nursing staff
  there was incomplete collection of data and patients dropped out which resulted in 77 total analyzed participants in this group
Arm/Group | Music Group | Midazolam Group
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/80
Other Adverse Events (participants affected / at risk) | 0/77 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/77/NCT03069677/Prot_SAP_000.pdf